CLINICAL TRIAL: NCT06208605
Title: Innovations in Personalizing Treatment for Eating Disorders Using Idiographic Methods and the Impact of Personalization on Psychological, Physical, and Sociodemographic Outcomes
Brief Title: Innovations in Personalizing Treatment Study
Acronym: T-NIPT-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cheri Levinson, Director, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#23.0529; 1DP2MH136495-01 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2024-01-17 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Eating Disorders
Keywords: Eating disorder; Treatment; Public Health; anorexia nervosa; bulimia nervosa; binge eating disorder; Other specified feeding and eating disorder; atypical anorexia nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdiagnostic Network Informed Personalized Treatment (Experimental): Participants will receive 1 session of education about the treatment after completing Phase I of the study (two weeks of ecological momentary assessment). Participants will then complete 10 sessions of personalized treatment for eating disorders based on their ecological momentary assessment surveys. Participants will complete one session of relapse prevention at the end.
  Interventions: Behavioral: Transdiagnostic Network Informed Personalized Treatment
- Cognitive Behavioral Therapy for Eating Disorders (Active Comparator): Participants will receive 1 session of education about the treatment after completing Phase I of the study (two weeks of ecological momentary assessment). Participants will then complete 10 sessions of Enhanced Cognitive Behavioral Therapy for Eating Disorders (CBT-E. Participants will complete one session of relapse prevention at the end.
  Interventions: Behavioral: Enhanced Cognitive Behavioral Therapy for Eating Disorders

INTERVENTIONS:
Behavioral: Transdiagnostic Network Informed Personalized Treatment — Idiographic network analysis is used to determine individuals' top central eating disorder symptoms. Participants then receive modules to address these specific symptoms.
  Other Names: Personalized Treatment
  Arms: Transdiagnostic Network Informed Personalized Treatment
Behavioral: Enhanced Cognitive Behavioral Therapy for Eating Disorders — Manualized CBT-E (Fairburn 2008) including regular eating, self-monitoring, and CBT modules implemented flexibly.
  Other Names: CBT-E
  Arms: Cognitive Behavioral Therapy for Eating Disorders

SUMMARY:
Eating disorders (EDs) are serious mental illness: someone dies of an ED every 52 minutes. EDs are highly related to a host of negative outcomes, including public health and individual disease burden, medical and psychological comorbidities, and social determinants of health (SDOH). Treatment response for EDs are suboptimal; there are no evidence-based treatment for adults with anorexia nervosa (AN) or Other Specified Feeding or Eating Disorder (OSFED) and only 50% of adults respond to current evidence based treatments. There are no precision treatments, nor any treatments that consider social context, in existence. Personalized treatments for EDs, that consider social contexts, are urgently needed to improve treatment response and minimize the suffering associated with these illnesses. The investigators' overall goal, extending upon their past work, is to create a treatment personalized based on idiographic (or one person) models (termed Transdiagnostic Network Informed Personalized Treatment for EDs; T-NIPT-ED). The investigators will carry out a two-phase study to systematically characterize individual mechanisms of treatment (Phase I: N=900) and then test the efficacy of each treatment module (Phase II: N=240 drawn from Phase I) compared to the current gold-standard treatment (Cognitive Behavioral Therapy Enhanced: CBT-E). The study goals are to (1) characterize the prevalence of T-NIPT-ED precision treatment mechanisms and medical and psychological comorbidities (e.g., obesity; depression), individual disease burden (e.g., disability), SDOH (e.g., food insecurity), and public health outcomes (e.g., service utilization) specific to these mechanisms, (2) identify if personalized target mechanisms improve when matched to evidence-based treatment modules of T-NIPT-ED and (3) test if change in T-NIPT-ED is associated with improved outcomes (vs CBT-E), including ED outcomes, comorbidities, disease burden, and public health outcomes and if these outcomes are moderated by SDOH. These goals will ultimately lead to the very first precision treatment for ED and can be extended to additional psychiatric illnesses. The proposed research uses highly innovative methods; intensive longitudinal data collected with mobile technology is combined with state-of-the art idiographic modeling methods to deliver a virtual, personalized treatment. This proposal integrates assessment of broad (e.g., SDOH; public health burden) and specific (e.g., ED symptoms) outcomes, to ensure that social context can be integrated into personalization. The proposed research has high clinical impact. Ultimately, this proposal will lead directly to the creation and dissemination of an evidence-based individually-personalized treatment for EDs, as well as will serve as an exemplar for precision treatment development across the entire field of psychiatry.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of any active eating disorder except ARFID
* Ages 18-65

Exclusion Criteria:

* Active Suicidality
* Active Mania
* Active psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-01-21 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Eating disorder symptoms | Up to 18 weeks
  Eating Disorder Examination Questionnaire 6.0 (EDE-Q) will be used to measure change in eating disorder symptoms. The EDEQ has a minimum global score of 0 and a maximum global score of 132. Higher scores indicate more severe eating pathology.
Clinical impairment | Up to 18 weeks
  The Clinical Impairment Assessment (CIA) will be used to measure change in severity of psychosocial impairment. The CIA has a minimum score of 0 and a maximum score of 48, with higher scores indicating higher levels of impairment.

SECONDARY OUTCOMES:
Psychological comorbidities using Structured Clinical Interview for DSM-5 (SCID-5) | Up to 18 weeks
  The investigators will be assessing psychological comorbidities using the SCID-5. The SCID-5 is a semi-structured interview used to arrive at DSM-5 diagnoses. Participants will complete the ED, anxiety, depression, mania, psychosis, and suicide modules.
Medical comorbidities using the Health Utilization and Medical Comorbidities | Up to 18 weeks
  The investigators will measure medical comorbidities (e.g., obesity) using the Health Utilization and Medical Comorbidities measure. This measure does not have a score but rather asks questions about different types of healthcare services and medical conditions and whether the participant has/has used them.
Health service utilization using the Health Utilization and Medical Comorbidities | Up to 18 weeks
  The investigators will measure health service utilization using the Health Utilization and Medical Comorbidities measure. This measure does not have a score but rather asks questions about different types of healthcare services and medical conditions and whether the participant has/has used them.

CONTACTS AND LOCATIONS:
Overall Officials: Cheri A Levinson, PhD, Principal Investigator — University of Louisville
Locations (1):
- Eating Anxiety Laboratory and Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levinson CA, Williams BM, Christian C, Hunt RA, Keshishian AC, Brosof LC, Vanzhula IA, Davis GG, Brown ML, Bridges-Curry Z, Sandoval-Araujo LE, Ralph-Nearman C. Personalizing eating disorder treatment using idiographic models: An open series trial. J Consult Clin Psychol. 2023 Jan;91(1):14-28. doi: 10.1037/ccp0000785. PMID 36729494
- [Background] Borsboom D, Cramer AO. Network analysis: an integrative approach to the structure of psychopathology. Annu Rev Clin Psychol. 2013;9:91-121. doi: 10.1146/annurev-clinpsy-050212-185608. PMID 23537483
- [Background] Levinson CA, Hunt RA, Keshishian AC, Brown ML, Vanzhula I, Christian C, Brosof LC, Williams BM. Using individual networks to identify treatment targets for eating disorder treatment: a proof-of-concept study and initial data. J Eat Disord. 2021 Nov 4;9(1):147. doi: 10.1186/s40337-021-00504-7. PMID 34736538